CLINICAL TRIAL: NCT01473108
Title: Study to Investigate the Effectiveness of Different Single Oral Doses of BAY94-8862 on Natriuresis After Administration of 0.5 mg Fludrocortisone (Astonin H®) With 50 mg Eplerenone (Inspra®) as Active Control in Healthy Male Subjects in a Randomized, Single-blind, Placebo-controlled, Combined 3-fold Crossover and Parallel-group Design
Brief Title: Study to Investigate the Natriuretic Effects, Safety, Tolerability and Pharmacokinetics of BAY94-8862
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 13786; 2010-018500-90 (EudraCT Number)
Record Dates: First submitted 2011-08-18; First posted 2011-11-17 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Clinical Pharmacology
Keywords: Healthy volunteers, proof-of-concept trial, PK and PD
MeSH Terms: interventions — finerenone; Eplerenone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Finerenone (20 mg solution) (Experimental): 3-fold crossover of single dose 20 mg BAY 94-8862 solution, placebo and 50 mg eplerenone. The challenge drug fludrocortisone was given 2 h prior to administration of BAY 94-8862, eplerenone, and placebo.
  Interventions: Drug: Finerenone (BAY 94-8862) PEG solution; Drug: Eplerenone (Inspra®); Drug: Placebo
- Finerenone (10 mg solution) (Experimental): 3-fold crossover of single dose 10 mg BAY 94-8862 solution, placebo and 50 mg eplerenone. The challenge drug fludrocortisone was given 2 h prior to administration of BAY 94-8862, eplerenone, and placebo.
  Interventions: Drug: Finerenone (BAY 94-8862) PEG solution; Drug: Eplerenone (Inspra®); Drug: Placebo
- Finerenone (5 mg solution) (Experimental): 3-fold crossover of single dose 5 mg BAY 94-8862 solution, placebo and 50 mg eplerenone. The challenge drug fludrocortisone was given 2 h prior to administration of BAY 94-8862, eplerenone, and placebo.
  Interventions: Drug: Finerenone (BAY 94-8862) PEG solution; Drug: Eplerenone (Inspra®); Drug: Placebo
- Finerenone (20 mg as tablets) (Experimental): 3-fold crossover of single dose 20 mg BAY 94-8862 as 2 x 10 mg tablet, placebo and 50 mg eplerenone. The challenge drug fludrocortisone was given 2 h prior to administration of BAY 94-8862, eplerenone, and placebo.
  Interventions: Drug: Finerenone (BAY 94-8862) immediate release tablet; Drug: Eplerenone (Inspra®); Drug: Placebo
- Finerenone (2.5 mg solution) (Experimental): 3-fold crossover of single dose 2.5 mg BAY 94-8862 solution, placebo and 50 mg eplerenone. The challenge drug fludrocortisone was given 2 h prior to administration of BAY 94-8862, eplerenone, and placebo.
  Interventions: Drug: Finerenone (BAY 94-8862) PEG solution; Drug: Eplerenone (Inspra®); Drug: Placebo

INTERVENTIONS:
Drug: Finerenone (BAY 94-8862) PEG solution — 2.5, 5, 10, 20 mg polyethylene glycol (PEG) solution of BAY 94-8862
  Arms: Finerenone (10 mg solution); Finerenone (2.5 mg solution); Finerenone (20 mg solution); Finerenone (5 mg solution)
Drug: Finerenone (BAY 94-8862) immediate release tablet — 20 mg BAY 94-8862 administered as 2 x 10 mg IR tablets
  Arms: Finerenone (20 mg as tablets)
Drug: Eplerenone (Inspra®) — Single oral dose of 50 mg eplerenone
Drug: Placebo — Matching placebo (solution/tablet) corresponding to BAY 94-8862 dose in respective dose step

SUMMARY:
Pharmacodynamics, pharmacokinetics, safety, and tolerability will be investigated in this single dose study. In 5 treatment groups, different dosages of BAY94-8862 will be given in healthy male subjects.

DETAILED DESCRIPTION:
Clinical pharmacology

ELIGIBILITY:
Inclusion Criteria:

* Healthy male white subjects
* 18 to 46 years of age
* Body mass index (BMI): 18 - 29.9 kg/m²

Exclusion Criteria:

* Clinically relevant findings in medical history or in the physical examination
* Systolic blood pressure below 100 or above 140 mmHg
* Diastolic blood pressure below 50 or above 90 mmHg
* Heart rate below 45 or above 95 beats / min

Ages: 18 Years to 46 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2010-03-29 (Actual); Primary Completion 2010-11-30 (Actual); Study Completion 2011-05-17 (Actual)

PRIMARY OUTCOMES:
Log10 (10*urinary Na+/K+ ratio) (Parameter for natriuresis) | Up to 26 hours post-dose
AUC (Area under the concentration vs time curve from zero to infinity after single (first) dose for both BAY 94-8862 and eplerenone) | Up to 60 hours after administration
Cmax (Maximum observed drug concentration in measured matrix after single dose administration for both BAY 94-8862 and eplerenone) | Up to 60 hours after administration

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/